CLINICAL TRIAL: NCT04439500
Title: Preventing Cognitive and Functional Decline Among Seniors at Risk-Effects of Online Training Aimed at Increasing Participation in Everyday Life During a Pandemic.
Brief Title: Effects of Online Training Aimed at Increasing Participation in Everyday Life During a Pandemic (SCD Online).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Dr. Deirdre Dawson, Rotman Research Institute, Baycrest, Baycrest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REB1738- sub-study
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Subjective Cognitive Decline
Keywords: Age-related cognitive changes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real World Strategy Training (Experimental): Group intervention including education and strategy training to manage everyday functional difficulties.
  Interventions: Behavioral: Real World Strategy Training
- Psychosocial Education (Active Comparator): Group sessions including education on brain health.
  Interventions: Behavioral: Brain Education

INTERVENTIONS:
Behavioral: Real World Strategy Training — The key features of the protocol are: i. Participants are actively engaged in selecting their treatment goals. The research clinician will work with the participants to identify five specific, measurable real-world goals using a standardized semi-structured interview, the Canadian Occupational Performance Measure. Three of these will be training goals, two will not be trained but evaluated post-intervention for evidence of generalization and transfer to non-trained tasks; ii. A global problem solving approach is used (Goal- Plan- Do- Check). Participants are guided by the trainer to apply this strategy to their goals.
  Arms: Real World Strategy Training
Behavioral: Brain Education — The active comparator uses an information-based format and is designed to engage participants without providing any specific training techniques or strategies. During weekly sessions, participants will receive factual information on brain structure and function, age-related cognitive changes, and general brain health issues and will spend time doing non-specific cognitive exercises including crossword and Sodoku puzzles. Homework will consist of reading assignments related to the session topics.
  Arms: Psychosocial Education

SUMMARY:
This study evaluates the efficacy of Real-World Strategy Training (RWST) compared to a psycho-education workshop for improving everyday life performance in older adults with subjective cognitive decline (SCD). Participants will be randomly assigned to receive one of these approaches. Additionally, this study will provide insight into the benefits of the program while people are not able to meet in person during a pandemic.

DETAILED DESCRIPTION:
Evidence suggests that 25-50% of community-dwelling older adults report SCD and that these individuals have an elevated risk for developing Mild Cognitive Impairment and/or dementia. Many of these individuals report difficulties with complex activities of daily living.

RWST aims to reduce these difficulties in everyday life by providing a meta-cognitive training approach that compensates for age-related executive changes. The approach is provided within the context of individually identified everyday-life difficulties.

The psycho-education approach is a Brain-Health Workshop supplemented by intellectually stimulating activities such as doing Sudoku and/or word searches. This approach provides information people may use to inform health behaviour changes.

ELIGIBILITY:
Inclusion Criteria:

* Have access to high speed internet and a computer or mobile device with a webcam
* Have subjective cognitive complaints
* Be fluent in written and spoken English
* Able to self-identify areas of their everyday lives in which they would like to improve.

Exclusion Criteria:

* Diagnosis of neurological conditions (e.g. dementia, mild cognitive impairment, Parkinson's)
* Presence of severe depression
* Presence of substance abuse
* History of hospitalization for psychiatric reasons

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in improved performance (measured as total number of untrained goals improved to criterion) on the Canadian Occupational Performance Measure (COPM) immediately post-intervention. | Changes from baseline to post-intervention at 10 weeks
  The COPM is a standardized semi-structure interview in which participants identify everyday life difficulties (defined as things they need to or want to do). These issues are converted to goals with performance rated on a 10-point Likert-type scale. Goals considered improved to criterion are those that have a 2 or more points increase on ratings.

SECONDARY OUTCOMES:
Improved performance on the Canadian Occupational Performance Measure (COPM) measured at three and six months post-intervention. | Three and six months post-intervention
  Same as outcome 1. Goals considered improved to criterion are those that have a 2 or more points increase on ratings.
Improved satisfaction with performance on trained and untrained goals identified using the COPM. | 10 weeks after baseline (after intervention), 3 months post-intervention, 6 months post-intervention
  Satisfaction with performance is measured on a 10-point Likert type scale using the Canadian Occupational Performance Measure. Goals considered improved to criterion are those that have a 2 or more points increase on ratings.
Changes on Social Support Survey Instrument (MOS-SSS) | Baseline, 10 weeks, 3 months post-intervention, 6 months post-intervention
  This 5-point likert type instrument measures participants' perceived availability of social support in various situations. The lowest possible score is 20 and highest possible is 100. Higher scores indicate better outcome.
Changes on DeJong Gierveld Loneliness Scale | Baseline, 10 weeks, 3 months post-intervention, 6 months post-intervention
  This scale measures loneliness and perceived social isolation. It will be administered to evaluate the impact of the intervention on participants' levels of self-isolation and loneliness. Lowest possible score is 0 and highest score is 6. Lower scores indicate better outcome.
Changes on Lubben Social Network Scale | Baseline, 10 weeks, 3 months post-intervention, 6 months post-intervention
  This 5-point likert type scale measures social isolation by measuring frequency, size, and closeness of contacts of the respondent's social network by assessing the perceived level of support they get from friends and families. Lowest possible score is 0 and highest possible score is 30. Higher scores indicate better outcome.
Change in health-related Quality of Life | Baseline, 10 weeks, 3 months post-intervention, 6 months post-intervention
  Health-related quality of life will be measured using the Short From Health Survey (SF-36). This survey includes the following sub scales (higher scores on each sub-scale indicate better outcome):
  Physical functioning with lowest possible score being 10 and highest 30; Role functioning with lowest possible score of 4 and highest 8; Bodily pain with lowest possible score of 2 and highest of 12; General health with lowest possible score of 5 and highest of 25; Vitality with lowest possible score of 4 and highest of 24; Social functioning with lowest possible score of 2 and highest of 10; Role-emotional with lowest possible score of 3 and highest of 6; Mental health with lowest possible score of 5 and highest of 30.

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Dawson, PhD, Principal Investigator — Rotman Research Institute, Baycrest Health Sciences
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada